CLINICAL TRIAL: NCT06550089
Title: A Pilot Study of High Or Low Dose pOstpartUm Oxytocin at the Time of Cesarean Birth (HOLDOUT Pilot)
Brief Title: High Or Low Dose pOstpartUm Oxytocin at the Time of Cesarean Birth
Acronym: HOLDOUT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study will be restarted at a later date
Sponsor: University of Chicago (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB24-0398
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-08

CONDITIONS: Postpartum Hemorrhage; Pregnancy Complications; Cesarean Section Complications
Keywords: oxytocin; cesarean delivery; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage; Pregnancy Complications | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High-dose oxytocin (Experimental): 900 mL/hr (54 units/hr) intravenously for the duration of the cesarean delivery
  Interventions: Drug: Oxytocin
- Low-dose oxytocin (Active Comparator): For unlabored cesarean births: 300 mL/hr (18 IU/hr), with a maximum rate of 900 mL/hr (54 units/hr) intravenously for the duration of the cesarean delivery
  For laboring cesarean births: 600 mL/hr (36 IU/hr), with a maximum rate of 900 mL/hr (54 units/hr) intravenously for the duration of the cesarean delivery
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin is a synthetic molecule used to reduce the likelihood of postpartum hemorrhage.

SUMMARY:
This is a study to investigate whether it is feasible to conduct a randomized controlled trial (RCT) of a high dose of oxytocin versus the standard low-dose oxytocin. Further the investigators, aim to assess whether there are differences in health outcomes between both arms of the study.

DETAILED DESCRIPTION:
Due to risks of postpartum hemorrhage, defined by the American College of Obstetricians and Gynecologists, as an estimated or quantitative blood loss of greater than 1000 milliliters, uterotonics, or medications aimed at increasing uterine tone and reducing blood loss at the time of birth, are commonly administered. Based on a Cochrane network meta-analysis, most organizations endorse the administration of 10 international units (IU) of oxytocin during delivery. However, the World Health Organization specifies that during a cesarean birth, the 10 IU should be administered using a bolus dose and an infusion, though an optimal infusion rate has yet to be agreed upon.

The use of a higher rate of oxytocin may confer a reduction in overall blood loss and subsequent maternal health outcomes (e.g., postoperative anemia, hypotension) and healthcare resource utilization (e.g., need for additional uterotonics and surgical procedures to control bleeding, administration of blood products). However, it is unknown whether it is feasible to conduct a randomized controlled trial to investigate the use of high (i.e., oxytocin rate of 900 mL/hr immediately after the delivery of the placenta) versus low-dose oxytocin (i.e., 300 mL/hr for planned cesarean births or 600 mL/hr for intrapartum cesarean births).

ELIGIBILITY:
Inclusion criteria.

* Age 18 or greater
* English or Spanish speaking
* Individuals undergoing a scheduled or unscheduled cesarean delivery

Exclusion criteria

* Patient on therapeutic anticoagulation
* Patient with hypertensive disorder of pregnancy or chronic hypertension
* Patient with preexisting bleeding disorder
* Patient with preexisting cardiac disease
* Patient with severe asthma, defined as the need for two or more agents for disease control, or bronchospasm
* Patient undergoing planned cesarean hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Screen failure rate | Within 8 hours prior to cesarean delivery
  Number of individuals who are eligible for the study but do not consent to participate
Fidelity rate | Within 8 hours prior to cesarean delivery
  Frequency of fidelity to the trial
Trial retention rate | Up to 6 weeks after cesarean delivery
  Frequency of participant completion of all study visits
Acceptability of the intervention | Up to 6 weeks after cesarean delivery
  Frequency of acceptability of the intervention by both participants and their providers

SECONDARY OUTCOMES:
Maternal flushing | During and up to 6 hours after cesarean delivery
Maternal hypotension | During and up to 6 hours after cesarean delivery
  Mean arterial blood pressure less than 65 mmHg
Maternal nausea/vomiting | During and up to 6 hours after cesarean delivery
Myocardial ischemia | During and up to 24 hours after cesarean delivery
Cardiac arrhythmia | During and up to 24 hours after cesarean delivery
Quantitative blood loss greater than 1 liter | Within 24 hours after cesarean delivery
Need for blood product transfusion, inclusive of type and number of blood products transfused | Within 4 days after cesarean delivery
Frequency of increase in oxytocin rate in low-dose arm | During and up to 6 hours after cesarean delivery
Additional use of uterotonics and/or tranexamic acid | During and up to 24 hours after cesarean delivery
Placement of intrauterine balloon tamponade or suction device | During and up to 24 hours after cesarean delivery
Surgical management of hemorrhage, inclusive of hysterectomy | During and up to 24 hours after cesarean delivery
Intensive care unit admission | During and up to 24 hours after cesarean delivery
Maternal death | During and up to 6 weeks after cesarean delivery
Readmission to the hospital or reoperation | Up to 6 weeks after cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Premkumar, MD, PhD, Principal Investigator — University of Chicago; Anna Palatnik, MD, Principal Investigator — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared by the us, the investigators, upon request by other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code